CLINICAL TRIAL: NCT06628661
Title: Ten-Year Outcomes of Operable Solitary Hepatocellular Carcinoma Patients: Impact of Tumor Size Over 6.5 Cm and Microvascular Invasion
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMRPG3N0051; MOHW112-CMAP-M-113-000006-D (Other: The Ministry of Health and Welfare, Taiwan)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma (HCC); Solitary Mass
Keywords: Hepatocellular carcinoma; Solitary tumor; Operable; Survival analysis; Tumor size; Microvacular invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Solitary HCC larger than 6.5 cm without mVI: Operable solitary HCC larger than 6.5 cm without mVI
  Interventions: Procedure: Surgery for HCC larger than 6.5 cm
- Solitary HCC larger than 2 cm with mVI: Operable solitary HCC larger than 2 cm with mVI
  Interventions: Procedure: Surgery for HCC larger than 2 cm

INTERVENTIONS:
Procedure: Surgery for HCC larger than 6.5 cm — Surgery for HCC larger than 6.5 cm without mVI
  Groups: Solitary HCC larger than 6.5 cm without mVI
Procedure: Surgery for HCC larger than 2 cm — Surgery for HCC larger than 2 cm with mVI
  Groups: Solitary HCC larger than 2 cm with mVI

SUMMARY:
The goal of this study is to evaualte the impact of tumor size and microvascular invasion among patients with solitary hepatocellualr carcinoma and post operation. The main questions it aims to answer are:

Does the tumor size have more impact on the survival and recurrence than microvascular invasion among solitary operable hepatocellular carcinoma patients?

Researchers will retrospectively analyze the prospectively collected clinical database during January 2022 and December 2019 to see whether tumor size more than 6.5 cm or microvascular invasion.

The solitary operable hepatocellular carcinoma patients would be classified based on the status of microvascular invasion and tumor size, and the outcome would be evaluated among different sub-populations of the feasible subjects.

DETAILED DESCRIPTION:
Data source The study utilized the Chang Gung Research Database (CGRD), an extensive repository of electronic medical records maintained by Chang Gung Memorial Hospital (CGMH) across multiple medical centers and hospitals in Taiwan. Established for administrative and insurance purposes, the CGRD includes comprehensive data on patient demographics, diagnoses, treatments, and outcomes. It covers a significant portion of Taiwan's medical services, with detailed records on outpatient, emergency, and inpatient visits. Notably, the CGRD also includes a cancer registry with thorough documentation of diagnoses, staging, treatment modalities, recurrence, and mortality data. All data in cancer registry database were curated manually and make this information highly reliable1. Diagnoses are coded using the International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) before 2016 and International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) thereafter, with all cancer registry entries manually verified for accuracy. This makes the CGRD an invaluable resource for clinical research. The CGRD's extensive coverage of Taiwan's medical landscape, including a significant proportion of both inpatient and outpatient services (20% of all cancer patients' data and about 34% outpatient information in Taiwan), underscores its utility as an excellent data source for robust clinical research. Previous studies have elaborated on the CGRD's structure and content, reinforcing its role as a key resource for healthcare studies.

Study design and population The study initially included all incident HCC patients from January 2002 to December 2018 by using ICD-9-CM codes 155 and ICD-10-CM codes C22. To ensure the population to be analyzed, several exclusion criteria were applied. Patients who did not receive any treatment after diagnosis were excluded to avoid confounding survival outcomes. Age was another critical factor; patients younger than 18 or older than 80 years were excluded to eliminate potential age-related biases in survival analysis. Additionally, patients with missing tumor size were excluded, as tumor size is a crucial variable in assessing prognosis and treatment decisions. Errors in survival or recurrence status or date were also excluded to maintain data integrity. Lastly, patients deemed non-operable were excluded to focus on those who could potentially benefit from surgical intervention. Furthermore, patients who did not fall into the pT1N0M0 or pT2N0M0 staging categories were excluded to ensure only early-stage patients were enrolled. The remaining patients were then divided into two groups based on their stage, in which subjects would be separated by TNM staging pT1N0M0 (solitary HCC) and pT2N0M0 (solitary HCC with mVi or multiple HCCs with none size < 5 cm). Within the pT1N0M0 group, patients who died within 30 days post-surgery were excluded to avoid perioperative mortality bias. Additionally, patients with a tumor size of ≤ 2cm were excluded to focus on more clinically significant tumors. Two subgroups, subjects with tumor size > 2cm and ≤ 6.5cm and > 6.5cm, were further obtained according to our previous report that 6.5 cm would be the cut-off value of pT1 subjects with different prognosis. For the pT2N0M0 group, similar exclusions were made for patients who died within 30 days post-surgery and for errors in the Child score. This group was further categorized into solitary tumor with microvascular invasion (mVI) and multiple tumors with none smaller than 5cm. Also, tumor size 6.5 cm was used to classify subjects with solitary tumor with mVi. The outcomes were compared among different groups of enrolled subjects to realize the associations between operation outcomes and HCC with mVi and tumor size over or below 6.5 cm among solitary HCC patients. This study, approved by the Institutional Review Board of the Chang Gung Medical Foundation, leverages the CGRD's rich data repository to conduct a retrospective cohort analysis (IRB No.: 202300142B0).

ELIGIBILITY:
Inclusion Criteria:

* Operable solitary hepatocellular carcinoma

Exclusion Criteria:

* Not pT1N0M0 or pT2N0M0
* Missing tumor size
* Errors in survival/recurrence dates or status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population would include different groups of enrolled subjects to realize the associations between operation outcomes and HCC with microvascular invasions and tumor size over or below 6.5 cm among solitary HCC patients.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
10-year overall survival | From enrollment to the end date of 10 years or the mortality occurs.
  10-year overall survival of different cohorts

SECONDARY OUTCOMES:
10-year disease-free survival | From enrollment to the end date of 10 years or the mortality or recurrence occur.
  10-year disease-free survival of different cohorts
10-year liver-specific survival | From enrollment to the end date of 10 years or the mortality due to liver condiiton occurs.
  10-year liver-specific survival of different cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
The IPD would be available upon adequte request.

REFERENCES:
- [Background] Lee CW, Yu MC, Wang CC, Lee WC, Tsai HI, Kuan FC, Chen CW, Hsieh YC, Chen HY. Liver resection for hepatocellular carcinoma larger than 10 cm: A multi-institution long-term observational study. World J Gastrointest Surg. 2021 May 27;13(5):476-492. doi: 10.4240/wjgs.v13.i5.476. PMID 34122737
- [Background] Lee CW, Tsai HI, Yu MC, Wang CC, Lee WC, Yeh TS, Yeh CN, Lin CY, Kuo T, Chen HY. A proposal for T1 subclassification in hepatocellular carcinoma: reappraisal of the AJCC 8th edition. Hepatol Int. 2022 Dec;16(6):1353-1367. doi: 10.1007/s12072-022-10422-8. Epub 2022 Sep 28. PMID 36169915